CLINICAL TRIAL: NCT04466085
Title: A Randomized, Blinded, Placebo-controlled Trial to Evaluate the Immunogenicity and Safety of a Recombinant New Coronavirus Vaccine (CHO Cell) With Different Doses and Different Immunization Procedures in Healthy People Aged 18 to 59 Years
Brief Title: Clinical Study of Recombinant Novel Coronavirus Vaccine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCV-Ⅱ-healthy
Record Dates: First submitted 2020-07-08; First posted 2020-07-10 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Coronavirus
Keywords: NOVID-19
MeSH Terms: conditions — Coronavirus Infections | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Population I (Experimental): In population I, there were 150 subjects who injected with 2 doses of low-dose test vaccine into the deltoid muscle of the upper arm according to the 0 and 1 month immunization schedule.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cell) low-dose group
- Population II (Experimental): In population II, there were 150 subjects who injected with 2 doses of high-dose test vaccine in the upper arm deltoid muscle according to the 0 and 1 month immunization schedule.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cells) high-dose group
- Population Ⅲ (Placebo Comparator): In population Ⅲ, there were 150 subjects who injected with 2 doses of placebo in the upper arm deltoid muscle according to the 0 and 1 month immunization schedule.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cells) placebo group
- Population Ⅳ (Experimental): In population Ⅳ, there were 150 subjects who injected with 3 doses of low-dose test vaccine in the upper arm deltoid muscle according to the 0, 1, and 2 month immunization schedule.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cell) low-dose group
- Population Ⅴ (Experimental): In population Ⅴ, there were 150 subjects who injected with 3 doses of high-dose test vaccine into the deltoid muscle of the upper arm according to the immunization schedule of 0, 1, and 2 months.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cells) high-dose group
- Population Ⅵ (Placebo Comparator): In Population Ⅵ, there were 150 subjects who injected with 3 doses of placebo into the deltoid muscle of the upper arm according to the immunization schedule of 0, 1, and 2 months.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cells) placebo group

INTERVENTIONS:
Biological: Recombinant new coronavirus vaccine (CHO cell) low-dose group — Intramuscular injection of deltoid muscle of upper armof 25μg/0.5ml/person doseRecombinant new coronavirus vaccine (CHO cells).
  Arms: Population I; Population Ⅳ
Biological: Recombinant new coronavirus vaccine (CHO cells) high-dose group — Intramuscular injection of deltoid muscle of upper armof 50μg/0.5ml/person doseRecombinant new coronavirus vaccine (CHO cells).
  Arms: Population II; Population Ⅴ
Biological: Recombinant new coronavirus vaccine (CHO cells) placebo group — Intramuscular injection of deltoid muscle of upper armof 0.5ml/person doseRecombinant new coronavirus vaccine (CHO cells).
  Arms: Population Ⅲ; Population Ⅵ

SUMMARY:
A total of 900 subjects are planned to be randomly divided into 2 doses of low-dose experimental vaccine group, 2 doses of high-dose experimental vaccine group, 2 doses of placebo group, 3 doses of low-dose experimental vaccine group, 3 doses of high-dose experimental vaccine group and 3 doses of placebo group, the sample size of each group was 150 cases.

DETAILED DESCRIPTION:
A total of 900 subjects are planned to be randomly divided into 2 doses of low-dose experimental vaccine group, 2 doses of high-dose experimental vaccine group, 2 doses of placebo group, 3 doses of low-dose experimental vaccine group, 3 doses of high-dose experimental vaccine group and 3 doses of placebo group, the sample size of each group was 150 cases.

Subjects in the 2 dose group were injected with 2 doses of test vaccine or placebo in the upper arm deltoid muscle according to the 0,1 month immunization program, and subjects in the 3 dose group were injected with 3 doses of test vaccine or placebo in the upper arm deltoid muscle according to the 0, 1, 2 month immunization program .

ELIGIBILITY:
Inclusion Criteria:

* Persons with full civil capacity aged 18-59 years (both included);
* The subjects themselves voluntarily agreed to participate in the study, and signed an informed consent form, and can provide valid identification; understand and comply with the requirements of the trial protocol;
* Body temperature under armpit <37.3℃;
* Female and male subjects of childbearing age agreed to take effective contraceptive measures during the study.

Exclusion Criteria:

* The vital signs and physical examination results of the population specified in the plan have clinical significance as determined by the clinician;
* A history of severe allergies to any component of the test vaccine, including aluminum preparations, such as: anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrosis (Arthus reaction), dyspnea, vascular neuropathy Edema, etc.; or any previous history of serious side effects after using any vaccine or drug;
* Those with a history of SARS and SARS-CoV-2 (meet any of the following: ① previous history of SARS and SARS-CoV-2 infection or morbidity; ② during the current SARS-CoV-2 epidemic, there are patients diagnosed/suspected with the new crown Contact history);
* Have taken antipyretics or painkillers within 24 hours before the first dose of vaccination;
* Within 14 days before the first dose of vaccination, subunit vaccines, inactivated vaccines, and live attenuated vaccines within 30 days;
* People with the following diseases: Acute febrile disease; Digestive diseases (eg, diarrhea, abdominal pain, vomiting, etc.) in the past 7 days; Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.; Congenital or Acquired immunodeficiency or a history of autoimmune diseases or treatment with immunomodulators within 6 months, such as hormones; or monoclonal antibodies; or thymosin; or interferon, etc.; however, topical medications (such as ointment, eye drops, Inhalation or nasal spray); known to be diagnosed with infectious diseases, such as: patients with tuberculosis, viral hepatitis and/or human immunodeficiency virus HIV positive or syphilis specific antibody positive; neurological disease or Neurodevelopmental dysplasia (eg, migraine, epilepsy, stroke, seizures in the last three years, encephalopathy, focal neurological deficit, Guillain-Barré syndrome, encephalomyelitis or transverse myelitis); history of psychiatric illness or family History; functional spleenlessness, and spleenlessness or splenectomy for any reason; severe chronic disease or disease in progress that cannot be controlled smoothly, such as diabetes, thyroid disease; severe liver and kidney disease; respiratory tract that currently requires daily medication Diseases (eg, chronic obstructive pulmonary disease [COPD], asthma) or any treatment that exacerbates respiratory diseases (eg, asthma exacerbations) within the last 5 years; has severe cardiovascular disease (eg, congestive heart failure, cardiomyopathy, Ischemic heart disease, arrhythmia, conduction block, myocardial infarction, pulmonary heart disease) or a history of myocarditis or pericarditis; with thrombocytopenia, any coagulopathy, or treatment with anticoagulants; tumor patients;
* Have received blood or blood-related products, including immunoglobulin, within 3 months; or plan to use it during the study;
* Women who are breastfeeding or pregnant (including a positive urine pregnancy test);
* Have used any research or unregistered product (medicine, vaccine, biological product or device) other than the research product within 3 months, or plan to use it during the research;
* The researchers believe that any disease or condition in the subject may put the subject at an unacceptable risk; the subject cannot meet the protocol requirements; and interfere with the assessment of vaccine response.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 900 (Actual)
Dates: Start 2020-07-12 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Neutralizing antibody positive conversion rate | 30 days after inoculation
  Neutralizing antibody positive conversion rate in the pre-immunization negative population 30 days after full vaccination

SECONDARY OUTCOMES:
Neutralizing antibody GMT, positive rate | 14 days after inoculation
  GMT and positive rate of neutralizing antibody 14 days after the first dose of pre-vaccination people
Neutralizing antibody GMT, positive conversion rate/positive rate | 14 days after inoculation
  GMT, positive conversion rate/positive rate of neutralizing antibodies 14 days after full vaccination in the pre-vaccination population
Neutralizing antibody GMT | 30 days after inoculation
  Neutralizing antibody GMT 30 days after vaccination in pre-negative people
Neutralizing antibody GMT | 6th and 12th month after inoculation
  Neutralizing antibody GMT in the 6th and 12th month after the entire vaccination
Neutralizing antibody GMI, positive rate | 6th and 12th month after inoculation
  Neutralizing antibody GMI and positive rate at the 6th and 12th month of the entire vaccination
IL-2, IL-4, IL-5, IL-6 and IFN-γ levels | 4th day and 12 months after inoculation
  Levels of IL-2, IL-4, IL-5, IL-6 and IFN-γ on the 4th day and 12 months after the entire vaccination
Adverse events | 30 days after inoculation
  Adverse events 30 days after the first dose of vaccine to the entire exemption
Serious adverse event | 12 months after inoculation
  Serious adverse events from day 0 after vaccination to 12 months after the entire immunization

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincial Center for Disease Control and Prevention, Hunan, Changsha, China

REFERENCES:
- [Derived] Yang S, Li Y, Dai L, Wang J, He P, Li C, Fang X, Wang C, Zhao X, Huang E, Wu C, Zhong Z, Wang F, Duan X, Tian S, Wu L, Liu Y, Luo Y, Chen Z, Li F, Li J, Yu X, Ren H, Liu L, Meng S, Yan J, Hu Z, Gao L, Gao GF. Safety and immunogenicity of a recombinant tandem-repeat dimeric RBD-based protein subunit vaccine (ZF2001) against COVID-19 in adults: two randomised, double-blind, placebo-controlled, phase 1 and 2 trials. Lancet Infect Dis. 2021 Aug;21(8):1107-1119. doi: 10.1016/S1473-3099(21)00127-4. Epub 2021 Mar 24. PMID 33773111